CLINICAL TRIAL: NCT05143307
Title: Long-Term Follow-Up Study of HIV-1 Infected Adults Exiting a Parent Study Where EBT-101 Was Administered
Brief Title: Long-Term Follow-Up Study of HIV-1 Infected Adults Who Received EBT-101
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Excision BioTherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EBT-101-002
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: HIV-1-infection
Keywords: CRISPR; Gene Therapy; adeno-associated virus serotype 9 (AAV9)

STUDY DESIGN:
Intervention Model Description: Long term follow up of participants who received EBT-101
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Long Term Follow Up (Experimental): Participants who received EBT-101 in a parent study will undergo long term follow up
  Interventions: Biological: EBT-101

INTERVENTIONS:
Biological: EBT-101 — Long term follow up of participants who received EBT-101

SUMMARY:
Participants who receive EBT-101 in a parent protocol will be eligible to participate in this long-term follow-up (LTFU) study (EBT-101-002).

DETAILED DESCRIPTION:
Participants who receive EBT-101 in a parent protocol will be eligible to participate in this LTFU study (EBT-101-002). All participants will have follow-up visits every six months until Year 5 post EBT-101. Thereafter, all participants will have follow-up visits annually on the anniversary of EBT-101 administration until study completion at Year 15.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written, signed informed consent
* Participants who received the investigational study intervention EBT-101 in a parent study

Exclusion Criteria:

• Participants who did not receive EBT-101 in a parent study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2037-01 (Estimated); Study Completion 2037-04 (Estimated)

PRIMARY OUTCOMES:
Long-term safety of EBT-101 | 15 years
  Long-term safety of EBT-101 will be assessed based on incidence and severity of clinically significant adverse events (AEs) according to Division of AIDS (DAIDS) 2017 over 15 years

CONTACTS AND LOCATIONS:
Overall Officials: William Kennedy, MD, Study Director — Excision BioTherapeutics
Locations (3):
- United States (3):
  - Quest Clinical Research, San Francisco, California
  - Washington University, St Louis, Missouri
  - Cooper Health, Camden, New Jersey

IPD SHARING:
Plan to Share IPD: No